CLINICAL TRIAL: NCT04423757
Title: A Phase II 6-week, Randomized, Double-blinded, Placebo Controlled, Parallel Group Decentralised Clinical Trial to Evaluate Efficacy and Safety of Oral BI 1358894 in Patients With Major Depressive Disorder With Inadequate Response to Antidepressants
Brief Title: A Home-based Study Using Mobile Technology to Test Whether BI 1358894 is Effective in People With Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1402-0014
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1358894 (Experimental): 125 milligram (mg) BI 1358894 taken orally as three film-coated tablets (1x 25mg and 2x 50mg) once a day in the morning for six weeks.
  Interventions: Drug: BI 1358894
- Placebo (Placebo Comparator): Placebo matching BI 1358894 taken orally as three film-coated tablets once a day in the morning for six weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1358894 — 125 milligram (mg) BI 1358894 taken orally as three film-coated tablets (1x 25mg and 2x 50mg) once a day in the morning for six weeks.
  Arms: BI 1358894
Drug: Placebo — Placebo matching BI 1358894 taken orally as three film-coated tablets once a day in the morning for six weeks.
  Arms: Placebo

SUMMARY:
This is a home-based study in adults with depression. People who have been diagnosed with Major Depressive Disorder can participate in the study. Participants can take part if they are being treated for their depression but still have symptoms. The purpose of this study is to find out whether a medicine called BI 1358894 helps people with depression.

Participants are in the study for about 2 months and do not need to visit a study site during this time. All study visits are conducted at participant's home by a mobile study nurse, by videoconference, and by phone calls. Participants are put into 2 groups by chance. One group takes BI 1358894 tablets. The other group takes placebo tablets. Placebo tablets look like BI 1358894 tablets but do not contain any medicine.

The participants answer questions about the symptoms of their depression. We then compare the results between the BI 1358894 and placebo groups. The doctors and nurses also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Major Depressive Disorder, single episode or recurrent, as confirmed at the time of screening by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders v5 (DSM-5, SCID-5), with a duration of current depressive episode ≥ 8 weeks and ≤ 12 months at the time of screening visit.
* Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥ 22 at screening, as confirmed by a trained rater. In addition, trial participants must have a score of ≥ 3 on the Reported Sadness item on MADRS.
* A documented ongoing monotherapy treatment of ≥ 8 weeks at the screening visit, with a protocol specified SSRI or SNRI (refer to the ISF) at adequate dose (at least minimum effective dose as per prescribing information and as confirmed per detectable drug levels in the screening blood or urine sampling).
* Male and female participants, 18 to 65 years of age, both inclusively at the time of consent.
* Women of child-bearing potential (WOCBP)2 able and willing to use two methods of contraception, which include one highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1%, plus one barrier method.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Able to communicate well, and to understand and comply with trial requirements.

Exclusion Criteria:

* Per DSM-5, had ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder or MDD with psychotic features as assessed by the Structured Clinical Interview for DSM -5 (SCID-5) at the time of screening.
* Diagnosis of any other mental disorder (in addition to those as described in Exclusion Criterion #1) that was the primary focus of treatment within 6 months prior to screening or at baseline (as per clinical discretion of the investigator).
* Diagnosis with antisocial, paranoid, schizoid or schizotypal personality disorder as per DSM-5 criteria, at the time of screening visit. Any other personality disorder at screening visit that significantly affects current psychiatric status and likely to impact trial participation, as per the judgement of investigator.
* Diagnosis of a substance related disorder within 3 months prior to screening visit (with exception of caffeine and tobacco).
* History of seizure disorders, stroke, brain tumor or any other major neurological illness that can impact participation in the trial.
* History of 4 or more unsuccessful monotherapy treatments (at adequate dosage and duration, per local prescribing information of the product) with an approved antidepressant medication for the current ongoing major depressive episode. These include ongoing monotherapy treatment with a protocol specified SSRI or SNRI as described in Inclusion Criterion #3.
* Any suicidal behavior in the past 12 months prior to screening (per investigator judgement including an actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour).
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months prior to screening or at screening or baseline visit (i.e. active suicidal thought with method and intent but without specific plan, or active suicidal thought with method, intent and plan).
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Science 37, Inc., Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted as a decentralized clinical trial (DCT). It was a 6-week parallel-group, randomized, double-blinded, placebo-controlled Phase II trial in participants with Major Depressive Disorder (MDD) with inadequate response to ongoing treatment of an Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin and Norepinephrine Reuptake Inhibitor (SNRI).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 1358894 | Placebo
Started | 21 | 24
Treated | 20 | 23
Completed (Based on completion of protocol specified treatment.) | 18 | 23
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all subjects who were randomized and received at least one administration of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1358894 | Placebo | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.4) | 43.2 (13.0) | 42.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 17 | 21 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 18 | 20 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Montgomery-Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: Score on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS) evaluates core symptoms of depression. Nine of the items are based upon participant reports, and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). Total score is calculated by the sum of the individual items, the possible total score could range from 0 to 60 (0= normal with absence of symptoms, 60=severe depression). Baseline for MADRS is last measurement prior to treatment start.
  Score on a scale | 26.6 (6.6) | 28.4 (7.1) | 27.6 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score at Week 6
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) evaluates core symptoms of depression. Nine of the items are based upon participant reports, and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). Total score is calculated by the sum of the individual items, the possible total score could range from 0 to 60 (0= normal with absence of symptoms, 60=severe depression). The adjusted mean (SE) are based on a mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect.
Time Frame: Week 0 (baseline) and after 1, 2, 4 and 6 week(s) of treatment. Change from baseline at week 6 MMRM estimates are reported in the table below.
Population: Full Analysis Set (FAS): all subjects who were randomized and received at least one administration of study drug that have a baseline and at least one evaluable post-baseline on-treatment measurement for the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 20 | 23
Score on a scale | -9.98 (NA) — Adjusted standard error = 2.3 | -13.36 (NA) — Adjusted standard error = 2.0
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom; Test type: Other; p = 0.2796, Mixed Models Analysis; Adjusted mean difference = 3.38, 90% CI 2-sided [-1.81 to 8.56], Standard Error of Mean 3.1 — Difference calculated as BI - Placebo

2. Secondary Outcome: Number of Subjects With ≥ 50% MADRS Reduction From Baseline at Week 6
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) evaluates core symptoms of depression. Nine of the items are based upon participant reports, and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). Total score is calculated by the sum of the individual items, the possible total score could range from 0 to 60 (0= normal with absence of symptoms, 60=severe depression). Reported are the number of subjects with ≥ 50% MADRS reduction from baseline at Weeks 6. Percent reduction from baseline was calculated as (score at baseline - score at week 6) / score at baseline * 100.
Time Frame: Baseline (week 0) and after 6 weeks of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 20 | 23
Participants | 6 | 14
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; Logistic regression includes treatment as covariate; Test type: Other; p = 0.0468, Regression, Logistic; Odds Ratio (OR) = 0.276, 90% CI 2-sided [0.091 to 0.781] — For the calculation of the odds ratio Placebo is taken as reference

3. Secondary Outcome: Change From Baseline in State-Trait Anxiety Inventory (STAI) Scores at Week 6
Description: The State-Trait Anxiety Inventory (STAI) comprises separate self-report scales for measuring state and trait anxiety. The S-Anxiety scale consists of twenty statements that evaluate how respondents feel "right now, at this moment." The T-Anxiety scale consists of twenty statements that assess how people generally feel. Scores for both the S-Anxiety and the T-Anxiety scales can vary from a minimum of 20 to a maximum of 80. Higher scores indicate greater anxiety.
  Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS): all subjects who were randomized and received at least one administration of study drug that have a baseline and at least one evaluable post-baseline on-treatment measurement for the primary endpoint. One subject in the BI 1358894 arm missed the baseline assessment for STAI and was excluded from this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 19 | 23
Score on a scale
  S-Anxiety scale | -9.10 (NA) — Adjusted standard error = 2.6 | -10.45 (NA) — Adjusted standard error = 2.3
  T-Anxiety scale | -8.70 (NA) — Adjusted standard error = 2.3 | -12.24 (NA) — Adjusted standard error = 2.0
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; S-Anxiety scale - Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom; Test type: Other; p = 0.6980, Mixed Models Analysis; Adjusted mean difference = 1.35, 90% CI 2-sided [-4.47 to 7.17], Standard Error of Mean 3.5 — Difference calculated as BI - Placebo
Statistical Analysis 2: Comparison: BI 1358894 vs Placebo; T-Anxiety scale - Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom; Test type: Other; p = 0.2589, Mixed Models Analysis; Adjusted mean difference = 3.54, 90% CI 2-sided [-1.67 to 8.76], Standard Error of Mean 3.1 — Difference calculated as BI - Placebo

4. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) Score at Week 6
Description: The CGI-S rating scale measures the clinician's impression of the severity of illness exhibited, taking into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 1 (best) to 7 (worst). Considering total clinical experience with the depression population, a participant is assessed on severity of illness at the time of rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. MMRM with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 20 | 23
Score on a scale | -1.14 (NA) — Adjusted standard error = 0.3 | -1.65 (NA) — Adjusted standard error = 0.3
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1863, Mixed Models Analysis; Adjusted mean difference = 0.51, 90% CI 2-sided [-0.13 to 1.15], Standard Error of Mean 0.4 — Difference calculated as BI - Placebo

5. Secondary Outcome: Change From Baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) Total Score at Week 6
Description: The SMDDS is a 16-item, patient-reported outcome (PRO) measure developed to capture the core symptoms of MDD. The SMDDS uses a recall of "over the past 7 days" and participants respond to each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"). In calculating the total score, two of the items (item 11 and 12) are first combined, with the highest score across the two items selected for use in the total score calculation. Total score is then calculated by the sum of the individual 15 items, the total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology. Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 19 | 23
Score on a scale | -13.56 (NA) — Adjusted standard error = 2.3 | -14.21 (NA) — Adjusted standard error = 2.0
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8326, Mixed Models Analysis; Adjusted mean difference = 0.65, 90% CI 2-sided [-4.46 to 5.76], Standard Error of Mean 3.1 — Difference calculated as BI - Placebo

6. Secondary Outcome: Change From Baseline in Patient Global Impression Severity Scale (PGI-S) Score at Week 6
Description: The PGI-S was used to measure the patient's impression of the severity of their illness. It is a single item 4-point scale that asks patients to rate the severity of their illness.
  The PGI-S question states "Please choose the response below that best describes the overall severity of your depression symptoms over the past week."
  1. None
  2. Mild
  3. Moderate
  4. Severe
  Mixed effects model for repeated measures (MMRM) with fixed effects of treatment, visit, treatment by visit interaction, baseline, and baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 11 | 14
Score on a scale | -0.37 (NA) — Adjusted standard error = 0.3 | -0.60 (NA) — Adjusted standard error = 0.2
Statistical Analysis 1: Comparison: BI 1358894 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5567, Mixed Models Analysis; Adjusted mean difference = 0.23, 90% CI 2-sided [-0.43 to 0.89], Standard Error of Mean 0.4 — Difference calculated as BI - Placebo

7. Secondary Outcome: Patient Global Impression of Change Scale (PGI-C) Score at Week 6
Description: The PGI-C is a one-time assessment at the end of treatment (EoT) to measure the patient's impression of the how their illness has changed over time. It is a single item 7-item scale that asks patients to rate the overall change since the start of treatment.
  The PGI-C question states "Please choose the response below that best describes the overall change in your depression symptoms since you started taking the study medication."
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: After 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 1358894 | Placebo
Number analyzed (Participants) | 20 | 23
Score on a scale | 2.8 (1.1) | 2.8 (1.7)

ADVERSE EVENTS:
Time Frame: From the date of first treatment administration till the date of the last treatment administration + Residual effect period, up to 70 days.
Description: Treated Set (TS): all subjects who were randomized and received at least one administration of study drug.
Arm/Group | BI 1358894 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/23
Other Adverse Events (participants affected / at risk) | 14/20 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1358894 (N=20) | Placebo (N=23)
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1358894 (N=20) | Placebo (N=23)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 5 | 2
Feeling abnormal (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 6 | 3
Somnolence (Nervous system disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hot flush (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Results should be interpreted in a descriptive manner since the trial was terminated early and the specified number of patients required for the analyses was not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04423757/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT04423757/SAP_001.pdf